CLINICAL TRIAL: NCT00818662
Title: A Randomized, Double-Blind, Placebo-Controlled, Two Dose Arm, Parallel Study of the Safety and Effectiveness of Immune Globulin Intravenous (Human), 10% (IGIV, 10%) for the Treatment of Mild-to-Moderate Alzheimer´s Disease
Brief Title: A Phase 3 Study Evaluating Safety and Effectiveness of Immune Globulin Intravenous (IGIV 10%) for the Treatment of Mild-to-Moderate Alzheimer´s Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 160701
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer´s Disease
Keywords: Alzheimer´s; Dementia; Dementia of Alzheimer Type; Immunoglobulins; Gammaglobulins; Immune Globulin Intravenous (IGIV); Intravenous Immune Globulin (IVIG); Antibodies; Amyloid; Immunotherapy
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — gamma-Globulins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IGIV, 10% 400mg/kg (Experimental): Immune Globulin Intravenous (Human), 10% (IGIV, 10%)
  Interventions: Biological: Immune Globulin Intravenous (Human), 10% (IGIV, 10%) 400 mg/kg
- IGIV, 10% 200mg/kg (Experimental): Immune Globulin Intravenous (Human), 10% (IGIV, 10%)
  Interventions: Biological: Immune Globulin Intravenous (Human), 10% (IGIV, 10%) 200 mg/kg
- Human Albumin 0.25% Solution - 4 mL/kg (Placebo Comparator): 0.25% human albumin solution infused at 4 mL/kg/2weeks
  Interventions: Biological: Placebo solution: Human Albumin 0.25% - 4 mL/kg
- Human Albumin 0.25% Solution - 2 mL/kg (Placebo Comparator): 0.25% human albumin solution infused at 2 mL/kg/2weeks
  Interventions: Biological: Placebo solution: Human Albumin 0.25% - 2 mL/kg

INTERVENTIONS:
Biological: Immune Globulin Intravenous (Human), 10% (IGIV, 10%) 400 mg/kg — 400 mg/kg bodyweight every 2 weeks for 70 weeks
  Other Names: Gammagard Liquid; KIOVIG
  Arms: IGIV, 10% 400mg/kg
Biological: Immune Globulin Intravenous (Human), 10% (IGIV, 10%) 200 mg/kg — 200 mg/kg bodyweight every 2 weeks for 70 weeks
  Other Names: Gammagard Liquid
  Arms: IGIV, 10% 200mg/kg
Biological: Placebo solution: Human Albumin 0.25% - 4 mL/kg — Placebo solution: 0.25% human albumin solution infused at 4 mL/kg/2weeks for 70 weeks
  Arms: Human Albumin 0.25% Solution - 4 mL/kg
Biological: Placebo solution: Human Albumin 0.25% - 2 mL/kg — Placebo solution: 0.25% human albumin solution infused at 2 mL/kg/2weeks for 70 weeks
  Arms: Human Albumin 0.25% Solution - 2 mL/kg

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of 2 doses of Immune Globulin Intravenous (IGIV), 10% administered every 2 weeks as an intravenous (IV) infusion compared with placebo in participants with mild to moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Study visits: Each participant will be tested at the investigational site, and if qualified, will be treated intravenously (through a vein) every two weeks for 70 weeks (approximately 18 months). The first three infusions must be done at the site, but if the infusions are well tolerated, subsequent infusions may be done by a qualified healthcare provider in the home or other suitable location. Each participant must return to the site every 3 months for evaluation of cognition as well as blood tests and scans of the brain.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent - participant (or participant´s legally acceptable representative) and caregiver who are willing and able to participate for the duration of the study
* Diagnosis of probable Alzheimer´s Disease (AD)
* Dementia of mild to moderate severity defined as mini-mental state examination (MMSE) 16-26 inclusive at the time of screening
* Neuroimaging (computed tomography [CT] or MRI) performed after symptom onset consistent with AD diagnosis
* Ability to comply with testing and infusion regimen, including fluency in English or Spanish, adequate corrected visual acuity and hearing ability
* On stable doses of regulatory authority approved AD medication(s) for at least 3 months prior to screening. These medications must be continued throughout this study.
* If receiving psychoactive medications (e.g. antidepressants other than monoamine oxidase inhibitors (MAOIs) and most tricyclics, antipsychotics, anxiolytics, anticonvulsants, mood stabilizers, etc), must be on stable doses for at least 6 weeks prior to screening

Main Exclusion Criteria (Reasons why it might not be appropriate to participate):

* Any other forms of dementia
* Medical issues that might increase the risk of treatment with IGIV, 10%, such as:

  1. Significant problems with blood pressure, heart disease, clotting disorders, strokes or recent heart attacks
  2. Evidence of current bleeding in the brain by MRI
  3. Serious problems with the liver or kidneys
  4. Allergies to blood products
* Medical issues that might interfere with the evaluation of the treatment of dementia or might make dementia worse, such as:

  1. Diabetes
  2. Recent treatment with chemotherapy or immune suppression
  3. The recent use of other investigational drugs, especially antibody therapy for AD
  4. Severe headaches or psychiatric problems

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2008-12-19 (Actual); Primary Completion 2012-12-10 (Actual); Study Completion 2012-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- United States (37):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Irvine, California
  - La Jolla, California
  - Los Angeles, California
  - National City, California
  - Orange, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Miami Beach, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Burlington, Massachusetts
  - Paw Paw, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Liverpool, New York
  - New York, New York
  - Rochester, New York
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - North Charleston, South Carolina
  - Franklin, Tennessee
  - Dallas, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin
- Canada (4):
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Background] Relkin N, Gessert D, Stokes K, Adamiak B, Ngo LY, Thomas R, Gelmont D, Aisen P. The Gammaglobulin Alzheimer Partnership Study (GAP): Design, screening, enrollment and futility analysis results. Alzheimer's & Dementia: The Journal of the Alzheimer's Association 8[4 Suppl], P456. 2012.
- [Background] Ngo L, Adamiak B, Gelmont D. A confirmatory phase 3 randomized, double-blind, placebo-controlled study of the safety and effectiveness of immune globulin intravenous (human), 10% solution (Gammagard Liquid/Kiovig) for the treatment of mild to moderate Alzheimer's Disease. Poster Presentation: Alzheimer's Association International Conference on Alzheimer's Disease (ICAD), Paris, France July 16-21 2011.
- [Derived] Relkin NR, Thomas RG, Rissman RA, Brewer JB, Rafii MS, van Dyck CH, Jack CR, Sano M, Knopman DS, Raman R, Szabo P, Gelmont DM, Fritsch S, Aisen PS; Alzheimer's Disease Cooperative Study. A phase 3 trial of IV immunoglobulin for Alzheimer disease. Neurology. 2017 May 2;88(18):1768-1775. doi: 10.1212/WNL.0000000000003904. Epub 2017 Apr 5. PMID 28381506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the U.S., and Canada, at 45 study sites. The first participant was enrolled in December 2008.
Pre-assignment Details: 702 participants were enrolled; 308 were screen failures; 4 were discontinued before randomization; and 7 were withdrawn after randomization, but prior to receiving investigational product. Therefore 383 participants were randomized.
Groups:
- IGIV, 10% 400mg/kg: Immune Globulin Intravenous (Human), 10% (IGIV, 10%) Immune Globulin Intravenous (Human), 10% (IGIV, 10%) : 400 mg/kg bodyweight every 2 weeks for 70 weeks
- IGIV, 10% 200mg/kg: Immune Globulin Intravenous (Human), 10% (IGIV, 10%) Immune Globulin Intravenous (Human), 10% (IGIV, 10%) : 200 mg/kg bodyweight every 2 weeks for 70 weeks
- Placebo 4 mL/kg: 0.25% human albumin solution infused at 4 mL/kg/2weeks Placebo solution: 4 mL/kg : 0.25% human albumin solution infused at 4 mL/kg/2weeks for 70 weeks
- Placebo 2 mL/kg: 0.25% human albumin solution infused at 2 mL/kg/2weeks Placebo solution: 2 mL/kg : 0.25% human albumin solution infused at 2 mL/kg/2weeks for 70 weeks
Period: Overall Study
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 4 mL/kg | Placebo 2 mL/kg
Started | 127 | 135 | 58 | 63
Completed | 104 | 102 | 49 | 47
Not Completed | 23 | 33 | 9 | 16
Not completed — Adverse Event | 5 | 14 | 4 | 3
Not completed — Withdrawal by Subject | 5 | 4 | 2 | 2
Not completed — Death | 1 | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Unwilling or Unable to Participate | 4 | 6 | 2 | 4
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Requires a Prohibited Medication | 1 | 0 | 0 | 0
Not completed — Safety Risk | 1 | 1 | 0 | 1
Not completed — Study Partner Unwilling or Unable | 3 | 2 | 1 | 1
Not completed — Participant's health declined | 0 | 0 | 0 | 1
Not completed — Caregiver to pursue other treatment | 0 | 1 | 0 | 0
Not completed — Moving out of state | 0 | 0 | 0 | 1
Not completed — Declined move to another study site | 1 | 0 | 0 | 0
Not completed — Change in living situation | 0 | 0 | 0 | 1
Not completed — Study partner decision | 0 | 0 | 0 | 1
Not completed — Admitted to long term nursing care | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 4 mL/kg | Placebo 2 mL/kg | Total
Number analyzed (Participants) | 127 | 135 | 58 | 63 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (9.6) | 70.1 (8.3) | 70.3 (9.7) | 70.1 (10.3) | 70.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 74 | 33 | 33 | 209
  Male | 58 | 61 | 25 | 30 | 174
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 117 | 127 | 56 | 58 | 358
  Canada | 10 | 8 | 2 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 18 Months in the Alzheimer´s Disease Assessment Scale- Cognitive Subscale (ADAS-Cog)
Description: The ADAS-Cog is a validated psychometric instrument that evaluates memory (word recall, word recognition), attention, reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing letter in envelope) and constructional praxis (copying geometric designs). This test was administered by experienced raters certified by Alzheimer's Disease Cooperative Study (ADCS) at each site. Scores on the ADAS-Cog range from 0-70 with higher scores indicating greater impairment; hence increases from baseline reflect potential cognitive deterioration.
Time Frame: Baseline & 18 months
Population: Intent-to-Treat Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- IGIV, 10% 400mg/kg: Immune Globulin Intravenous (Human), 10% (IGIV, 10%) Immune Globulin Intravenous (Human), 10% (IGIV, 10%) : 400 mg/kg bodyweight every 2 weeks for 70 weeks Adverse Events That Occurred During or After Treatment
- IGIV, 10% 200mg/kg: Immune Globulin Intravenous (Human), 10% (IGIV, 10%) Immune Globulin Intravenous (Human), 10% (IGIV, 10%) : 200 mg/kg bodyweight every 2 weeks for 70 weeks Adverse Events That Occurred During or After Treatment
- Placebo 2 mL/kg or 4 mL/kg: All participants who received the 2 mL/kg or 4 mL/kg placebo solution Placebo solution: 2 mL/kg or 4 mL/kg : 0.25% human albumin solution infused every 2 weeks for 70 weeks Adverse Events That Occurred During or After Treatment
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 105 | 100 | 95
Scores on a scale | 7.4 (7.95) | 8.9 (8.20) | 8.4 (9.37)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.476, ANCOVA; Difference in least-square means = -0.8, 95% CI [-3.1 to 1.5] — Results combined from 100 imputations from estimates & standard errors from 100 ANCOVA results for fixed effect of treatment, E4 allele of apolipoprotein E carrier status, & continuous covariates age at baseline, baseline ADAS-Cog & education level
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.530, ANCOVA; Difference in least-square means = 0.7, 95% CI [-1.6 to 3.0] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline at 18 Months in Alzheimer´s Disease Cooperative Study-Activities of Daily Living (ADCS-ADL)
Description: The ADCS-ADL scale is a validated tool to assess instrumental and basic activities of daily living based on a 23 item structured interview of the caregiver or qualified study partner. Scores on the ADCS-ADL range from 0-78 with lower scores indicating greater impairment; hence decreases from baseline reflect potential functional deterioration.
Time Frame: Baseline & 18 Months
Population: Intent-to-Treat Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo 2 mL/kg or 4 mL/kg: All participants who received the 2 mL/kg or 4 mL/kg placebo solution Placebo solution: 2 mL/kg or 4 mL/kg : 0.25% human albumin solution infused every 2 weeks for 70 weeks
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 104 | 102 | 95
Scores on a scale | -11.4 (10.49) | -12.4 (11.41) | -11.4 (12.19)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.812, ANCOVA; Difference in least-square means = 0.4, 95% CI [-2.9 to 3.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.602, ANCOVA; Difference in least-square means = -0.9, 95% CI [-4.3 to 2.5] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline at 9 Months in the Alzheimer´s Disease Assessment Scale- Cognitive Subscale (ADAS-Cog)
Description: as for outcome 1
Time Frame: Baseline & 9 months
Population: Intent-to-Treat Analysis Set with both baseline and month 9 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 114 | 114 | 106
Scores on a scale | 2.7 (5.20) | 4.5 (6.16) | 3.5 (6.44)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.368, ANCOVA; Difference in least-square means = -0.7, 95% CI [-2.3 to 0.8] — Estimated within a ANCOVA model accounting for the fixed effect of treatment, E4 allele of apolipoprotein E carrier status, and for the continuous covariates age at baseline, baseline ADAS-Cog and education level (in years)
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.319, ANCOVA; Difference in least-square means = 0.8, 95% CI [-0.8 to 2.4] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline at 9 Months in Alzheimer´s Disease Cooperative Study-Activities of Daily Living (ADCS-ADL)
Description: as for outcome 2
Time Frame: Baseline & 9 Months
Population: Intent-to-Treat Analysis Set with both baseline and month 9 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 111 | 116 | 107
Scores on a scale | -5.4 (7.03) | -6.1 (8.13) | -5.8 (8.32)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.778, ANCOVA; Difference in least-square means = 0.3, 95% CI [-1.8 to 2.4] — Estimated within a ANCOVA model accounting for the fixed effect of treatment, E4 allele of apolipoprotein E carrier status, and for the continuous covariates age at baseline, baseline ADCS-ADL and education level (in years)
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.851, ANCOVA; Difference in least-square means = -0.2, 95% CI [-2.3 to 1.9] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline at 9 Months in Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) Assessment
Description: The ADCS-CGIC is a validated categorical measure of change in a participant's clinical condition between baseline and follow-up visits; it is used to assess global clinical status. The ADCS CGIC score is based on direct examination of the participant and an interview of the caregiver. The rater should refer to the baseline ADCS-CGIC worksheets in making a rating. A skilled and experienced clinician who is blinded to treatment assignment rates the participant on a 7-point Likert scale, ranging from 1 (marked improvement) to 7 (marked worsening). 1= Very much better 2= Much better 3= A little better 4= Same 5= A little worse 6= Much worse 7= Very much worse
Time Frame: Baseline & 9 Months
Population: Intent-to-Treat Analysis Set with both baseline and month 9 assessments.
Measure: Number; unit: participants
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 114 | 114 | 104
participants
  Month 9: Very much better (1) | 0 | 0 | 0
  Month 9: Much better (2) | 2 | 1 | 1
  Month 9: A little better (3) | 7 | 3 | 7
  Month 9: Same (4) | 33 | 33 | 36
  Month 9: A little worse (5) | 52 | 56 | 48
  Month 9: Much worse (6) | 19 | 18 | 12
  Month 9: Very much worse (7) | 1 | 3 | 0
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.306, Mixed Models Analysis; Difference in least-square means = 0.1, 95% CI [-0.1 to 0.3]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.028, Mixed Models Analysis; Difference in least-square means = 0.3, 95% CI [0.0 to 0.5]

6. Secondary Outcome: Change From Baseline at 18 Months in Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) Assessment
Description: as for outcome 5
Time Frame: Baseline & 18 Months
Population: Intent-to-Treat Analysis Set with both baseline and month 18 assessments.
Measure: Number; unit: participants
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 105 | 101 | 92
participants
  Month 18: Very much better (1) | 0 | 0 | 0
  Month 18: Much better (2) | 1 | 2 | 1
  Month 18: A little better (3) | 6 | 1 | 3
  Month 18: Same (4) | 15 | 15 | 16
  Month 18: A little worse (5) | 44 | 43 | 36
  Month 18: Much worse (6) | 32 | 33 | 32
  Month 18: Very much worse (7) | 7 | 7 | 4
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.660, Mixed Models Analysis; Difference in least-square means = -0.1, 95% CI [-0.3 to 0.2]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.766, Mixed Models Analysis; Difference in least-square means = 0.0, 95% CI [-0.2 to 0.3]

7. Secondary Outcome: Change From Baseline at 18 Months in the Modified Mini-Mental State Examination (3MS) Examination
Description: The 3MS is a comprehensive validated instrument that provides a 100 point composite rating for spatial and temporal orientation, verbal recall, simple attention, working memory, naming, repetition, comprehension, writing and constructional abilities. Scores range from 0 to 100 with lower values indicating greater impairment.
Time Frame: Baseline & 18 months
Population: Intent-to-Treat Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 103 | 102 | 91
Scores on a scale | -12.1 (13.12) | -15.3 (12.76) | -13.5 (10.95)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.206, ANCOVA; Difference in least-square means = 1.9, 95% CI [-1.0 to 4.8]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.331, ANCOVA; Difference in least-square means = -1.4, 95% CI [-4.3 to 1.5]

8. Secondary Outcome: Change From Baseline at 18 Months in the Neuropsychiatric Inventory (NPI) Assessment
Description: The NPI is a validated instrument used to assess behavioral psychopathology in AD; it evaluates the frequency and severity of 12 neuropsychiatric features including delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, aberrant motor activity, sleep and night-time behavior change, and appetite and eating change. The NPI total score ranged 0-144, with higher scores indicating greater impairment.
Time Frame: Baseline & 18 months
Population: Intent-to-Treat Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 104 | 102 | 94
Scores on a scale | 3.7 (12.93) | 4.9 (13.30) | 2.4 (10.77)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.640, ANCOVA; Difference in least-square means = 0.7, 95% CI [-2.1 to 3.4]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.075, ANCOVA; Difference in least-square means = 2.5, 95% CI [-0.3 to 5.3]

9. Secondary Outcome: Change From Baseline at 18 Months in the Logsdon Quality of Life in Alzheimer's Disease (QOL-AD) Assessment- Participant Response
Description: The QOL AD is a validated, 13-item instrument developed specifically for individuals with dementia. The assessment rates the participant's quality of life for physical, emotional, interpersonal, and environmental domains. The QOL-AD total score ranged 13-52. Lower scores on the QOL AD are associated with a lower quality of life.
Time Frame: Baseline & 18 months
Population: Intent-to-Treat Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 99 | 99 | 86
Scores on a scale | -0.5 (5.34) | -0.7 (4.40) | -1.5 (5.20)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.093, ANCOVA; Difference in least-square means = 1.1, 95% CI [-0.2 to 2.3]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.094, ANCOVA; Difference in least-square means = 1.1, 95% CI [-0.2 to 2.3]

10. Secondary Outcome: Change From Baseline at 18 Months in the Logsdon Quality of Life in Alzheimer's Disease (QOL-AD) Assessment- Caregiver Response
Description: as for outcome 9
Time Frame: Baseline & 18 months
Population: Intent-to-Treat Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 99 | 99 | 92
Scores on a scale | -3.0 (4.97) | -2.5 (5.17) | -1.6 (5.12)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs IGIV, 10% 200mg/kg; Test type: Superiority or Other; p = 0.096, ANCOVA; Difference in least-square means = -1.1, 95% CI [-2.3 to 0.2]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.123, ANCOVA; Difference in least-square means = -1.0, 95% CI [-2.2 to 0.3]

11. Secondary Outcome: Change From Baseline at 18 Months in the Adjunct Neuropsychological Testing: Wechsler Adult Intelligence Scale- Revised (WAIS-R) Digit Span Forward
Description: This test assesses working memory and attention, the rater asks the participant to repeat single-digit number sequences of increasing length, which are read aloud by the rater (in forward or backward order). Two trials are presented for each sequence length, and the test is ended when the participant misses both trials at a given sequence length. The WAIS-R score ranged from 0-14. Results are presented as total number correct; therefore, lower numbers represent greater impairment.
Time Frame: Baseline & 18 months
Population: Per-Protocol Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 97 | 93 | 88
correct responses | -0.8 (2.00) | -1.2 (2.21) | -1.1 (1.81)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.167, ANCOVA; Difference in least-square means = 0.4, 95% CI [-0.2 to 1.0]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.998, ANCOVA; Difference in least-square means = -0.0, 95% CI [-0.6 to 0.6]

12. Secondary Outcome: Change From Baseline at 18 Months in the Adjunct Neuropsychological Testing: Wechsler Adult Intelligence Scale- Revised (WAIS-R) Digit Span Backward
Description: as for outcome 11
Time Frame: Baseline & 18 months
Population: Per-Protocol Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 94 | 89 | 86
correct responses | -0.8 (1.95) | -1.2 (1.88) | -1.2 (1.79)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.173, ANCOVA; Difference in least-square means = 0.4, 95% CI [-0.2 to 0.9]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.744, ANCOVA; Difference in least-square means = 0.1, 95% CI [-0.4 to 0.6]

13. Secondary Outcome: Change From Baseline at 18 Months in the Adjunct Neuropsychological Testing: FAS Verbal Fluency
Description: In the FAS assessment of phenomic verbal fluency, participants are given 1 minute each to name as many words as they can that begin with a specified letter (F, A, S). To receive credit, words must be verifiable in a dictionary, cannot be proper nouns, and cannot be the same word or variations of the same word (e.g., the same word with a different ending, such as 'acts,' 'acted,' 'acting'). Results are presented as total number correct; therefore, lower numbers indicate greater impairment.
Time Frame: Baseline & 18 months
Population: Per-Protocol Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 96 | 91 | 85
correct responses | -4.7 (8.60) | -7.4 (9.00) | -6.3 (8.17)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.238, ANCOVA; Difference in least-square means = 1.5, 95% CI [-1.0 to 4.0]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.400, ANCOVA; Difference in least-square means = -1.1, 95% CI [-3.6 to 1.4]

14. Secondary Outcome: Change From Baseline at 18 Months in the Adjunct Neuropsychological Testing: Wechsler Adult Intelligence Scale- Revised (WAIS-R) Digit Symbol Substitution
Description: WAIS-R digit symbol substitution test assesses attention, psychomotor speed, complex scanning, visual tracking, and immediate memory. This test consists of 4 rows each with 25 small blank squares; above each square is a number between 1 and 9. At the top is a 'key,' which pairs each number (1 through 9) with an unfamiliar symbol. The participant has 90 seconds to work as quickly as possible (left to right across the rows) to fill in each blank square with the appropriate symbol based on the number above the square. Results are presented as total number correct; therefore, lower numbers indicate greater impairment.
Time Frame: Baseline & 18 months
Population: Per-Protocol Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 80 | 63 | 67
correct responses | -6.8 (10.61) | -7.7 (9.67) | -6.2 (7.34)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.695, ANCOVA; Difference in least-square means = -0.6, 95% CI [-3.6 to 2.4]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.410, ANCOVA; Difference in least-square means = -1.3, 95% CI [-4.5 to 1.9]

15. Secondary Outcome: Change From Baseline at 18 Months in the Adjunct Neuropsychological Testing: Animals Category Fluency
Description: In this test, which assesses semantic verbal fluency, participants are given 1 minute to name as many items in the category "animals" as possible. To receive credit that word cannot be a mythical animal, but can be an animal species; breed; male, female, or infant name for a species (e.g., bull, cow, calf); in addition, names for birds, fish, reptiles, and insects receive credit. Results are presented as total number correct; therefore, lower numbers indicate greater impairment.
Time Frame: Baseline & 18 months
Population: Per-Protocol Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 97 | 92 | 87
correct responses | -2.8 (4.06) | -2.2 (6.84) | -2.7 (3.82)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.988, ANCOVA; Difference in least-square means = -0.0, 95% CI [-1.5 to 1.5]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.555, ANCOVA; Difference in least-square means = 0.4, 95% CI [-1.0 to 1.9]

16. Secondary Outcome: Change From Baseline at 18 Months in the Adjunct Neuropsychological Testing: Trail-Making Test (TMT), Part A
Description: This test, which has 2 parts, is used to assess processing speed, visuomotor and perceptual scanning skills, and executive function. In Part A, 25 circles each containing a number between 1 and 25 are randomly placed on a sheet of paper, and the participant is asked to draw a line as quickly as possible between each circle in ascending numerical order. In Part B, 25 circles are again randomly placed on a sheet of paper; however, in this test 13 of the circles contain the numbers 1 through 13, and the remaining 12 circles contain the letters A through L. In this test, the participant must draw a line as quickly as possible between the circles in alternating between numbers and letters in ascending order (e.g., 1 to A, A to 2, 2 to B,…). Total values for TMT Part A range between 0 and 150 seconds. Results are presented as time to complete; therefore, higher numbers indicate greater impairment.
Time Frame: Baseline & 18 months
Population: Per-Protocol Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 83 | 75 | 74
seconds | 21.6 (36.93) | 20.5 (30.61) | 21.3 (35.50)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.783, ANCOVA; Difference in least-square means = -1.5, 95% CI [-12.2 to 9.2]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.700, ANCOVA; Difference in least-square means = -2.1, 95% CI [-13.1 to 8.8]

17. Secondary Outcome: Change From Baseline at 18 Months in the Adjunct Neuropsychological Testing: Trail-Making Test (TMT), Part B
Description: This test, which has 2 parts, is used to assess processing speed, visuomotor and perceptual scanning skills, and executive function. In Part A, 25 circles each containing a number between 1 and 25 are randomly placed on a sheet of paper, and the participant is asked to draw a line as quickly as possible between each circle in ascending numerical order. In Part B, 25 circles are again randomly placed on a sheet of paper; however, in this test 13 of the circles contain the numbers 1 through 13, and the remaining 12 circles contain the letters A through L. In this test, the participant must draw a line as quickly as possible between the circles in alternating between numbers and letters in ascending order (e.g., 1 to A, A to 2, 2 to B,…). Total values for TMT Part B range between 0 and 300 seconds. Results are presented as time to complete; therefore, higher numbers indicate greater impairment.
Time Frame: Baseline & 18 months
Population: Per-Protocol Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 61 | 51 | 50
seconds | 13.0 (60.49) | 28.4 (65.01) | 31.9 (66.32)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.191, ANCOVA; Difference in least-square means = -15.2, 95% CI [-38.0 to 7.7]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.892, ANCOVA; Difference in least-square means = -1.6, 95% CI [-25.4 to 22.1]

18. Secondary Outcome: Change From Baseline at 18 Months in the Adjunct Neuropsychological Testing: Clock Drawing Test
Description: In this test, which assesses constructional ability, visuoperception, and executive functioning, the participant is given a blank sheet of paper and asked to draw the face of a clock showing the numbers and 2 hands set to 'ten after eleven.' Results are presented as score obtained (range 0 to 5, with 0 indicating the greatest impairment).
Time Frame: Baseline & 18 months
Population: Per-Protocol Analysis Set with both baseline and month 18 assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 94 | 90 | 85
Scores on a scale | -0.7 (1.27) | -0.7 (1.15) | -0.6 (1.17)
Statistical Analysis 1: Comparison: IGIV, 10% 400mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.588, ANCOVA; Difference in least-square means = -0.1, 95% CI [-0.4 to 0.2]
Statistical Analysis 2: Comparison: IGIV, 10% 200mg/kg vs Placebo 2 mL/kg or 4 mL/kg; Test type: Superiority or Other; p = 0.351, ANCOVA; Difference in least-square means = -0.2, 95% CI [-0.5 to 0.2]

19. Secondary Outcome: Number of Participants Experiencing Study Product-related Non-serious Adverse Events (Non-SAEs), by System Organ Class
Time Frame: Throughout the study period, approximately 4 years
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
participants
  Blood and Lymphatic System Disorders | 7 | 2 | 1
  Cardiac Disorders | 1 | 0 | 4
  Eye Disorders | 1 | 1 | 0
  Gastrointestinal Disorders | 10 | 13 | 7
  General Disorders & Administration Site Conditions | 22 | 32 | 13
  Immune System Disorders | 0 | 1 | 0
  Infections and Infestations | 1 | 1 | 1
  Injury, Poisoning, and Procedural Complications | 5 | 1 | 0
  Investigations | 15 | 16 | 13
  Metabolism and Nutrition Disorders | 0 | 1 | 0
  Musculoskeletal and Connective Tissue Disorders | 7 | 5 | 0
  Nervous System Disorders | 33 | 34 | 24
  Psychiatric Disorders | 5 | 6 | 2
  Reproductive System and Breast Disorders | 0 | 1 | 0
  Respiratory, Thoracic and Mediastinal Disorders | 3 | 4 | 4
  Skin and Subcutaneous Tissue Disorders | 26 | 20 | 9
  Vascular Disorders | 10 | 18 | 17

20. Secondary Outcome: Number of Participants Experiencing Study Product-related Serious Adverse Events (SAEs), by System Organ Class
Time Frame: Throughout the study period, approximately 4 years
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
participants
  Cardiac Disorders | 1 | 0 | 1
  General Disorders & Administration Site Conditions | 0 | 0 | 1
  Immune System Disorders | 0 | 1 | 0
  Investigations | 0 | 2 | 0
  Nervous System Disorders | 1 | 2 | 0
  Psychiatric Disorders | 0 | 1 | 0
  Respiratory, Thoracic and Mediastinal Disorders | 0 | 1 | 1
  Vascular Disorders | 0 | 0 | 2

21. Secondary Outcome: Number of Participants Experiencing Any Non-serious Adverse Events (Non-SAEs), by System Organ Class
Description: Related and unrelated non-SAEs
Time Frame: Throughout the study period, approximately 4 years
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
participants
  Blood and Lymphatic System Disorders | 13 | 7 | 5
  Cardiac Disorders | 3 | 11 | 15
  Ear and Labyrinth Disorders | 4 | 3 | 5
  Endocrine Disorders | 1 | 0 | 1
  Eye Disorders | 14 | 5 | 9
  Gastrointestinal Disorders | 47 | 51 | 36
  General Disorders & Administration Site Conditions | 57 | 66 | 52
  Immune System Disorders | 1 | 7 | 3
  Infections and Infestations | 40 | 46 | 57
  Injury, Poisoning, and Procedural Complications | 36 | 37 | 50
  Investigations | 37 | 48 | 30
  Metabolism and Nutrition Disorders | 14 | 15 | 16
  Musculoskeletal and Connective Tissue Disorders | 40 | 44 | 27
  Neoplasms, Benign, Malignant and Unspecified | 8 | 8 | 13
  Nervous System Disorders | 63 | 73 | 53
  Psychiatric Disorders | 41 | 49 | 49
  Renal and Urinary Disorders | 13 | 16 | 12
  Reproductive System and Breast Disorders | 5 | 4 | 3
  Respiratory, Thoracic and Mediastinal Disorders | 23 | 35 | 23
  Skin and Subcutaneous Tissue Disorders | 49 | 52 | 31
  Social Circumstances | 0 | 1 | 0
  Surgical and Medical Procedures | 8 | 6 | 8
  Vascular Disorders | 22 | 30 | 31

22. Secondary Outcome: Number of Participants Experiencing Any Serious Adverse Events (SAEs), by System Organ Class
Description: Related and unrelated SAEs
Time Frame: Throughout the study period, approximately 4 years
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
participants
  Blood and Lymphatic System Disorders | 2 | 0 | 1
  Cardiac Disorders | 5 | 3 | 3
  Ear and Labyrinth Disorders | 1 | 0 | 0
  Gastrointestinal Disorders | 5 | 1 | 1
  General Disorders & Administration Site Conditions | 2 | 4 | 2
  Hepatobiliary Disorders | 0 | 1 | 1
  Immune System Disorders | 0 | 1 | 0
  Infections and Infestations | 2 | 2 | 4
  Injury, Poisoning, and Procedural Complications | 3 | 2 | 2
  Investigations | 1 | 2 | 1
  Metabolism and Nutrition Disorders | 1 | 1 | 2
  Musculoskeletal and Connective Tissue Disorders | 2 | 3 | 0
  Neoplasms, Benign, Malignant and Unspecified | 0 | 3 | 3
  Nervous System Disorders | 3 | 6 | 5
  Psychiatric Disorders | 2 | 4 | 3
  Renal and Urinary Disorders | 0 | 1 | 1
  Respiratory, Thoracic and Mediastinal Disorders | 1 | 2 | 3
  Surgical and Medical Procedures | 0 | 1 | 1
  Vascular Disorders | 4 | 0 | 4

23. Secondary Outcome: Number of Infusions Temporally Associated With Non-serious Adverse Events (Non-SAEs) and/or Serious Adverse Events (SAEs)
Description: Refers to non-SAEs and/or SAEs occurring during infusion or within 72 hours of completion of infusion (regardless of causality)
Time Frame: During or within 72 hours of completion of an infusion
Population: Safety Analysis Set
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
Number analyzed (Infusions) | 3883 | 3954 | 3691
Infusions | 396 | 467 | 349

24. Secondary Outcome: Number of Infusions With Causally Associated Non-serious Adverse Events (Non-SAEs) and/or Serious Adverse Events (SAEs)
Description: Each adverse event (AE) that was considered related to investigational product (IP) was linked to the most recent infusion administered
Time Frame: Throughout the study period, approximately 4 years
Population: Safety Analysis Set
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
Number analyzed (Infusions) | 3883 | 3954 | 3691
Infusions | 225 | 265 | 172

25. Secondary Outcome: Number of Infusions Discontinued, Slowed, or Interrupted Due to an Adverse Event (AE)
Time Frame: Throughout each infusion period
Population: Safety Analysis Set
Measure: Number; unit: Adverse events
Units Other Than Participants: Infusions
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
Number analyzed (Infusions) | 3883 | 3954 | 3691
Adverse events | 48 | 28 | 36

26. Secondary Outcome: Number of Participants Experiencing a Clinically Significant Decrease in Hemoglobin (>1.5 g/dL) Between Consecutive Visits
Time Frame: Throughout the study period, approximately 4 years
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
participants | 31 | 24 | 16

27. Secondary Outcome: Number of Participants Experiencing a Clinically Significant Rash
Description: Participants requiring systemic therapy or discontinuation from further treatment
Time Frame: Throughout the study period, approximately 4 years
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Number analyzed (Participants) | 127 | 135 | 121
participants
  Rash requiring discontinuation from treatment | 3 | 2 | 0
  Rash requiring systemic therapy | 19 | 16 | 8

ADVERSE EVENTS:
Time Frame: Throughout the study period of approximately 4 years
Groups:
- Placebo 2 mL/kg or 4 mL/kg: All participants who received the 2 mL/kg or 4 mL/kg placebo solution Placebo solution: 2 mL/kg or 4 mL/kg : 0.25% human albumin solution infused every 2weeks for 70 weeks Adverse Events That Occurred During or After Treatment
Arm/Group | IGIV, 10% 400mg/kg | IGIV, 10% 200mg/kg | Placebo 2 mL/kg or 4 mL/kg
Serious Adverse Events (participants affected / at risk) | 21/127 | 32/135 | 26/121
Other Adverse Events (participants affected / at risk) | 112/127 | 118/135 | 103/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV, 10% 400mg/kg (N=127) | IGIV, 10% 200mg/kg (N=135) | Placebo 2 mL/kg or 4 mL/kg (N=121)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Microcytic Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (2)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic Hernia, Obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 2 (3) | 0 (0)
Multi-Organ Failure (General disorders) | 0 (0) | 2 (2) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Joint Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Normal Pressure Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Partial Seizures (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Radicular Pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 2 (3)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Unresponsive To Stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vasogenic Cerebral Oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Confusional State (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic Disorder Due To A General Medical Condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Inguinal Hernia Repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic Stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Orthostatic Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV, 10% 400mg/kg (N=127) | IGIV, 10% 200mg/kg (N=135) | Placebo 2 mL/kg or 4 mL/kg (N=121)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 3 (3) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 4 (4) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 18 (23) | 19 (24) | 15 (16)
Nausea (Gastrointestinal disorders) | 16 (24) | 11 (23) | 10 (16)
Vomiting (Gastrointestinal disorders) | 12 (16) | 6 (10) | 5 (6)
Chills (General disorders) | 10 (12) | 15 (33) | 3 (3)
Fatigue (General disorders) | 10 (11) | 13 (35) | 12 (28)
Gait Disturbance (General disorders) | 2 (2) | 10 (12) | 3 (3)
Infusion Site Extravasation (General disorders) | 23 (32) | 15 (18) | 21 (30)
Oedema Peripheral (General disorders) | 5 (5) | 7 (9) | 6 (7)
Pyrexia (General disorders) | 7 (8) | 7 (15) | 4 (4)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (10) | 9 (13)
Upper Respiratory Tract Infection (Infections and infestations) | 8 (9) | 8 (9) | 10 (11)
Urinary Tract Infection (Infections and infestations) | 12 (16) | 8 (10) | 15 (21)
Contusion (Injury, poisoning and procedural complications) | 9 (9) | 13 (17) | 10 (20)
Fall (Injury, poisoning and procedural complications) | 14 (20) | 16 (20) | 23 (31)
Laceration (Injury, poisoning and procedural complications) | 7 (9) | 5 (5) | 9 (10)
Blood Pressure Increased (Investigations) | 19 (65) | 12 (67) | 9 (49)
Weight Decreased (Investigations) | 2 (2) | 7 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 7 (7) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 11 (13) | 8 (8)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8 (11) | 4 (6) | 5 (5)
Cerebral Microhaemorrhage (Nervous system disorders) | 8 (9) | 1 (1) | 4 (5)
Dizziness (Nervous system disorders) | 16 (23) | 13 (16) | 12 (15)
Headache (Nervous system disorders) | 29 (114) | 34 (101) | 22 (65)
Tremor (Nervous system disorders) | 1 (1) | 12 (13) | 5 (5)
Agitation (Psychiatric disorders) | 9 (9) | 10 (10) | 10 (12)
Anxiety (Psychiatric disorders) | 9 (12) | 14 (16) | 10 (15)
Confusional State (Psychiatric disorders) | 5 (5) | 13 (19) | 4 (6)
Depression (Psychiatric disorders) | 14 (14) | 16 (18) | 19 (22)
Insomnia (Psychiatric disorders) | 1 (1) | 9 (10) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 13 (19) | 13 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 3 (3) | 3 (5)
Eczema (Skin and subcutaneous tissue disorders) | 7 (9) | 3 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 21 (27) | 19 (27) | 6 (10)
Hypertension (Vascular disorders) | 14 (27) | 18 (27) | 11 (22)
Hypotension (Vascular disorders) | 3 (3) | 6 (7) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication (by USCD) or 12 months after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥45 days prior to submission or communication. Baxter may request an additional delay of ≤45 days(e.g., for intellectual property protection)